CLINICAL TRIAL: NCT04706273
Title: GORE® VIABAHN® Endoprosthesis Post-Marketing Surveillance Study (JPS 16-03)
Status: Completed | Type: Observational
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Other Study IDs: JPS 16-03
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Results first posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2023-10

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- GORE® VIABAHN® Endoprosthesis: Participants with symptomatic peripheral arterial disease in superficial femoral artery lesions.
  Interventions: Device: GORE® VIABAHN® Endoprosthesis

INTERVENTIONS:
Device: GORE® VIABAHN® Endoprosthesis — Participants receiving the GORE® VIABAHN® Endoprosthesis

SUMMARY:
This study will confirm device efficacy and safety in the clinical setting after the launch of the GORE® VIABAHN® Endoprosthesis for the treatment of symptomatic peripheral arterial disease in the superficial femoral arteries.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic peripheral arterial disease in superficial femoral artery lesions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with symptomatic peripheral arterial disease in superficial femoral artery lesions in Japan
Sampling Method: Non-Probability Sample
Enrollment: 321 (Actual)
Dates: Start 2016-08-25 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2022-12-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kansai Rousai, Amagasaki, Hyōgo, Japan

REFERENCES:
- [Derived] Iida O, Ohki T, Soga Y, Suematsu N, Nakama T, Yamaoka T, Tobita K, Ichihashi S. Five-year outcomes of the GORE VIABAHN Endoprosthesis for the treatment of complex femoropopliteal lesions from a Japanese postmarket surveillance study. Vasc Med. 2024 Aug;29(4):416-423. doi: 10.1177/1358863X241233528. Epub 2024 Mar 27. PMID 38544413

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: limbs
Period: Overall Study
Arm/Group | GORE® VIABAHN® Endoprosthesis
Started | 321; 324 limbs
Completed | 136; 136 limbs
Not Completed | 185; 188 limbs
Not completed — Withdrawal by Subject | 27
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 42
Not completed — Death | 85
Not completed — Amputation that removes study device | 2
Not completed — Surgical bypass | 3
Not completed — Changing hospital | 23
Not completed — Unable to attend hospital | 2

BASELINE CHARACTERISTICS:
Arm/Group | GORE® VIABAHN® Endoprosthesis
Number analyzed (Participants) | 321
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 3 participants are missing age
  years
    number analyzed (Participants) | 318
    (all) | 73.9 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73
  Male | 248
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Japan | 321

OUTCOME MEASURES:

1. Primary Outcome: Primary Assisted Patency
Description: Primary assisted patency is defined as hemodynamic evidence of flow through a device that had not required a Target lesion revascularization to restore flow after total occlusion. Kaplan-Meier estimates created for each time point.
Time Frame: 12 and 24 months
Population: Participant limbs treated
Measure: Number (95% Confidence Interval); unit: probability
Units Other Than Participants: limbs
Arm/Group | GORE® VIABAHN® Endoprosthesis
Number analyzed (Participants) | 321
Number analyzed (limbs) | 324
probability
  12 months | 0.920 [0.880 to 0.946]
  24 months | 0.873 [0.826 to 0.908]

2. Primary Outcome: Freedom From Target Lesion Revascularization
Description: Revascularization for restenosis or occlusion of the target lesion. Kaplan-Meier estimates created for each time point.
Time Frame: 1, 12 and 24 months
Population: Participant limbs treated
Measure: Number (95% Confidence Interval); unit: probability
Units Other Than Participants: limbs
Arm/Group | GORE® VIABAHN® Endoprosthesis
Number analyzed (Participants) | 321
Number analyzed (limbs) | 324
probability
  1 Month | 0.997 [0.978 to 1.000]
  12 Months | 0.924 [0.887 to 0.949]
  24 Months | 0.844 [0.797 to 0.881]

3. Primary Outcome: Number of Participants With One or More Device- or Procedure-related Serious Adverse Events and Deficiencies
Description: The number and proportion of the subjects for whom the occurrence of serious adverse events were reported.
Time Frame: Procedure day, 1, 12, 24, 36, 48 and 60 months
Population: Participants must have been followed for at least as long as the start day identified for the time period. Participants that discontinued prior to the start day of the time period were not included in the number analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GORE® VIABAHN® Endoprosthesis
Number analyzed (Participants) | 321
Participants
  Procedure (Day 0) | 7
  1 Month (Days 0 through 37) | 11
  3 Months (Days 38 through 121): number analyzed (Participants) | 316
  3 Months (Days 38 through 121) | 3
  6 Months (Days 122 through 212): number analyzed (Participants) | 310
  6 Months (Days 122 through 212) | 9
  12 Months (Days 213 through 395): number analyzed (Participants) | 306
  12 Months (Days 213 through 395) | 17
  24 Months (Days 396 through 760): number analyzed (Participants) | 292
  24 Months (Days 396 through 760) | 20
  36 Months (Days 761 through 1277): number analyzed (Participants) | 268
  36 Months (Days 761 through 1277) | 13
  48 Months (Days 1278 through 1642): number analyzed (Participants) | 214
  48 Months (Days 1278 through 1642) | 7
  60 Months (Days 1643 through 1855): number analyzed (Participants) | 184
  60 Months (Days 1643 through 1855) | 2

4. Primary Outcome: Number of Participants With a Stent Fracture
Description: The number and proportion of stent fracture as assessed by Core lab
Time Frame: Month 12, 24, 36, 48 and 60
Population: Includes all subjects who had an x-ray to determine device stent fracture status at the reported corresponding follow-up time period.
Measure: Count of Participants; unit: Participants
Arm/Group | GORE® VIABAHN® Endoprosthesis
Number analyzed (Participants) | 321
Participants
  12 Months: number analyzed (Participants) | 280
  12 Months | 0
  24 Months: number analyzed (Participants) | 244
  24 Months | 0
  36 Months: number analyzed (Participants) | 192
  36 Months | 0
  48 Months: number analyzed (Participants) | 150
  48 Months | 0
  60 Months: number analyzed (Participants) | 122
  60 Months | 0

ADVERSE EVENTS:
Time Frame: 60 months (Days 0 through 1855)
Description: The post-market surveillance study was conducted in compliance with GPSP (Good Post-marketing Study Practice). All Serious Adverse Events regardless of their causal relationship with the study device are reported. However, non-serious events that are not related to the study device or procedure are rarely reported. All non-serious events reported were not in sufficient quantity to meet the reporting frequency threshold for Other Adverse Events.
Arm/Group | GORE® VIABAHN® Endoprosthesis
All-Cause Mortality (participants affected / at risk) | 85/321
Serious Adverse Events (participants affected / at risk) | 188/321
Other Adverse Events (participants affected / at risk) | 0/321
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GORE® VIABAHN® Endoprosthesis (N=321)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2)
Acute on chronic heart failure (Cardiac disorders) | 3 (3)
Angina pectoris (Cardiac disorders) | 3 (3)
Aortic valve stenosis (Cardiac disorders) | 3 (3)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrial fibrillation paroxysmal (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 5 (6)
Cardiac failure acute (Cardiac disorders) | 4 (4)
Cardiac failure aggravated (Cardiac disorders) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Cardiac valvulopathy (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 3 (5)
Ischaemic heart disease (Cardiac disorders) | 1 (1)
Left anterior descending coronary artery stenosis (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1)
Mesenteric arterial occlusion (Gastrointestinal disorders) | 1 (1)
Mesenteric artery stenosis (Gastrointestinal disorders) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Arterial stent occlusion (General disorders) | 1 (1)
Death (General disorders) | 12 (12)
Found dead (cause undetermined) (General disorders) | 1 (1)
In-stent arterial restenosis (General disorders) | 2 (4)
In-stent arterial stenosis (General disorders) | 7 (11)
In-stent coronary artery restenosis (General disorders) | 2 (2)
Inflammatory reaction (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Stent restenosis (General disorders) | 1 (1)
Sudden arrhythmic death syndrome (General disorders) | 1 (1)
Sudden death (General disorders) | 2 (2)
Vascular stent-graft occlusion (General disorders) | 5 (5)
Vascular stent-graft stenosis (General disorders) | 24 (29)
Vascular stent-graft thrombosis (General disorders) | 1 (1)
Vessel puncture site haematoma (General disorders) | 1 (1)
Vessel puncture site haemorrhage (General disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Contrast media allergy (Immune system disorders) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Endocarditis infective (Infections and infestations) | 1 (1)
Gangrene (Infections and infestations) | 4 (4)
Panperitonitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 10 (13)
Pneumonia aspiration (Infections and infestations) | 6 (6)
Pneumonia bacterial (Infections and infestations) | 2 (2)
Postoperative wound infection (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 2 (3)
Sepsis (Infections and infestations) | 2 (2)
Septic shock (Infections and infestations) | 1 (2)
Urinary tract infection (Infections and infestations) | 1 (2)
Vascular stent graft infection (Infections and infestations) | 1 (1)
Acute subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Arterial bypass occlusion (Injury, poisoning and procedural complications) | 3 (4)
Arterial bypass stenosis (Injury, poisoning and procedural complications) | 1 (2)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1)
Arterial restenosis (Injury, poisoning and procedural complications) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Coronary artery reocclusion (Injury, poisoning and procedural complications) | 1 (1)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1 (1)
Femoral artery pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Femoropopliteal artery bypass occlusion (Injury, poisoning and procedural complications) | 1 (2)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Plaque shift (Injury, poisoning and procedural complications) | 1 (1)
Popliteal artery pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Superficial femoral arterial restenosis (Injury, poisoning and procedural complications) | 3 (4)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Trochanteric femoral fracture (Injury, poisoning and procedural complications) | 1 (1)
Ankle brachial index decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Nutritional condition abnormal (Investigations) | 1 (1)
Geromarasmus (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Knee deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Advanced lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Brain tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carcinomatous peritonitis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Liver tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6)
Lung cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bilateral recurrent laryngeal nerve paralysis (Nervous system disorders) | 1 (1)
Cardioembolic stroke (Nervous system disorders) | 2 (2)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 6 (6)
Epileptiform fits NOS (Nervous system disorders) | 1 (1)
Internal carotid artery stenosis (Nervous system disorders) | 2 (2)
Lacunar infarction (Nervous system disorders) | 1 (1)
Device occlusion (Product Issues) | 45 (60)
Suicide (Psychiatric disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 (1)
Bilateral pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial pneumonia aggravated (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Digital ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Ischaemic leg ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Lower extremities ulcers of (Skin and subcutaneous tissue disorders) | 1 (1)
Leg amputation (Surgical and medical procedures) | 2 (2)
Peripheral artery stent insertion (Surgical and medical procedures) | 1 (1)
Abdominal aortic aneurysm (Vascular disorders) | 1 (1)
Aortic aneurysm rupture (Vascular disorders) | 2 (2)
Arterial occlusion (Vascular disorders) | 1 (1)
Arterial stenosis leg (Vascular disorders) | 2 (2)
Arteriosclerosis obliterans (Vascular disorders) | 1 (1)
Claudication (Vascular disorders) | 1 (1)
Critical limb ischaemia (Vascular disorders) | 2 (2)
Dialysis hypotension (Vascular disorders) | 1 (1)
Femoral arterial stenosis (Vascular disorders) | 3 (3)
Femoral artery occlusion (Vascular disorders) | 1 (1)
Iliac artery dissection (Vascular disorders) | 1 (1)
Iliac artery occlusion (Vascular disorders) | 1 (1)
Iliac artery stenosis (Vascular disorders) | 5 (5)
Intermittent claudication (Vascular disorders) | 1 (1)
Lower limb ischaemia (Vascular disorders) | 1 (1)
Obstructive arteriosclerosis of lower extremities (Vascular disorders) | 6 (8)
Peripheral embolism (Vascular disorders) | 2 (2)
Popliteal artery occlusion (Vascular disorders) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 3 (3)
Subclavian artery stenosis (Vascular disorders) | 2 (2)
Superficial femoral arterial stenosis (Vascular disorders) | 8 (10)
Superficial femoral artery occlusion (Vascular disorders) | 18 (18)
Thoracic aortic aneurysm (Vascular disorders) | 1 (1)
Tibial artery occlusion (Vascular disorders) | 2 (2)
Tibial artery stenosis (Vascular disorders) | 1 (1)
Vascular dissection (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI is required to obtain written permission from the Sponsor prior to publishing trial results.

DOCUMENTS (2):
  • Study Protocol (2016-06-07): https://cdn.clinicaltrials.gov/large-docs/73/NCT04706273/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT04706273/SAP_001.pdf